CLINICAL TRIAL: NCT05395949
Title: A Randomized Controlled Study of Conservative Treatment of Granulomatous Lobular Mastitis Combined With Psychiatric Disorders
Acronym: GLMwPD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Chair, Department of Thyroid and Breast Surgery, Zhongnan Hospital of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLMwPD
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Breast Diseases; Mastitis Granulomatous; Psychiatric Disorder
Keywords: granulomatous lobular mastitis ；Psychiatric Disorder；Steroid
MeSH Terms: conditions — Breast Diseases; Granulomatous Mastitis; Mental Disorders | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid combined with methotrexate (Experimental): Prednisone 30 mg/day, supplemented with calcium and omeprazole, and Prednisone were slowly reduced to 10 mg/day after symptoms were relieved, and combined with 7.5 mg/week MTX therapy.
  Interventions: Drug: conservative treatment
- Extensive lesion excision (No Intervention): Patients in the control group underwent wide local excision, make sure the margin is negative. Irrigation and mammoplasty were performed in the same way as in the observation group.

INTERVENTIONS:
Drug: conservative treatment — Prednisone 30 mg/day, supplemented with calcium and omeprazole, and Prednisone were slowly reduced to 10 mg/day after symptoms were relieved, and combined with 7.5 mg/week MTX therapy.
  Arms: Steroid combined with methotrexate

SUMMARY:
Granulomatous lobular mastitis (GLM) is a relatively rare chronic inflammatory disease of the breast in clinical practice. A small number of patients develop hyperprolactinemia during psychiatric drug treatment, and most of these patients are nulliparous. At present, there is no unified treatment mode at home and abroad, and surgery is generally the main treatment. GLM is a sterile inflammation, and glucocorticoids and methotrexate can effectively relieve clinical symptoms and even reach the standard of cure. In order to reduce the recurrence rate and protect the breast appearance as much as possible, we propose a conservative therapy. The purpose of this study was to compare this conservative therapy of granulomatous lobular mastitis with existing surgical treatment, and to compare the overall benefits of the two for patients with GLM. We aim to protect the breast appearance on the premise of low recurrence, improve the quality of life of GLM patients with psychiatric disorders .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with granulomatous lobular mastitis
* Patients with Psychiatric Disorders;
* Patients volunteered to participate in the study after informed consent.

Exclusion Criteria:

* Patients were diagnosed with mastitis with other definite etiology confirmed by pathology
* Patients in acute exacerbation of mental illness

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | Up to 1 years
  Inflammatory changes, mass, abscess or fistula formation, nodular erythema of the upper and lower extremities and joint pain occurred in the ipilateral breast within one year after surgery was defined as recurrence.
Breast appearance and cosmetic effect score | Up to 1 years
  Refer to Harris standard to evaluate postoperative cosmetic effect. Specify the breast appearance and cosmetic effect rating table.

SECONDARY OUTCOMES:
recovery time | Up to 2 years
  the timing of the disappearance of the symptoms including Inflammatory changes, mass, abscess or fistula formation, nodular erythema of the upper and lower extremities and joint pain occurred in the ipilateral breast

CONTACTS AND LOCATIONS:
Overall Officials: Gaosong Wu, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No